CLINICAL TRIAL: NCT03936075
Title: Guided Imagery & Music in Active Treatment for Gynecologic or Breast Cancer: An RCT Pilot
Brief Title: Guided Imagery & Music in Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aalborg University (Other)
Collaborators: Aretaieion University Hospital (Other); SONORA Organisation for Music Therapy and Research (Unknown)
Responsible Party: Principal Investigator, Evangelia Papanikolaou, Evangelia Papanikolaou, music therapist, Principal Investigator, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 62/19-06-18
Record Dates: First submitted 2019-04-29; First posted 2019-05-03 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Cancer, Breast; Cancer, Metastatic; Cancer Ovaries; Cancer Uterus Cervix
Keywords: receptive music therapy; Guided Imagery & Music (GIM); chemotherapy; radiotherapy; breast cancer; gynecologic cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Ovarian Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: two randomised groups, one intervention group and one placebo group
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): treatment with the provision of 6 individual sessions of the Guided Imagery and Music method as a psychological supportive intervention, and psychometric questionnaires collection
  Interventions: Behavioral: the Guided Imagery and Music method
- control (Placebo Comparator): standard care treatment with psychometric questionnaires collection and two individual counselling sessions, at baseline (week 1) and at the end (week 6)
  Interventions: Behavioral: standard care and verbal counselling

INTERVENTIONS:
Behavioral: the Guided Imagery and Music method — the method involves listening to the music while describing the experience to the therapist, any visual imagery that is evoked by the music, emotions, body sensations, thoughts or memories. after the music listening session, there is discussion upon making meaning of the experience and finding resources as potential coping skills
  Other Names: receptive music psychotherapy
  Arms: intervention
Behavioral: standard care and verbal counselling — the participants receive their usual cancer treatment and two individual counselling sessions
  Arms: control

SUMMARY:
This is an RCT pilot study to explore the potential effects of the Guided Imagery & Music method for women with breast or gynecologic cancer, during active treatment. The study explores the potential impact in quality of life parameters such as mood, fatigue, and hope.

DETAILED DESCRIPTION:
Guided Imagery and Music is a music-assisted psychotherapy method which has been used as a complementary, supportive psychosocial therapy in cancer care. However, its effects have never been explored during the period of active chemotherapy or radiotherapy treatment in various cancer populations, and especially gynecologic and breast cancer. This pilot study is an effort to explore the feasibility of the method to increase quality of life in this population by possibly reducing side-effects of treatment such as fatigue, improving mood, and building resilience as expressed through levels of hope.

ELIGIBILITY:
Inclusion Criteria:

* Speaking Greek
* receiving chemotherapy or radiotherapy treatment for breast or gynecologic cancer
* first occurrence or metastatic
* have an interest in engaging in creative psychotherapies through music

Exclusion Criteria:

* women with active psychosis or PTSD symptomatology
* women receiving other psychological support
* women too ill to participate according to doctors' instructions

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Profiles of Mood States (POMS) Brief version (adapted) | Baseline and up to 12 weeks (post-intervention)
  Brief version adapted in Greek. A 30-item scale designed to assess six different moods namely tension, anger, vigor, fatigue, depression, confusion. It requires to indicate mood state over the last week, with a single word, each item ranging from 0(not at all) to 4 (extremely). The questionnaire is a sum of its 6 sub scales (each addressing the aforementioned moods), with a total score from 0 to 120. Lower scores indicate better mood states.

SECONDARY OUTCOMES:
Herth Hope Index | Baseline and up to 12 weeks (post-intervention)
  A 12-item Likert-format instrument assessing current levels of hope from 1(strongly disagree) to 4 (strongly agree). It consists of three sub scales, examining interconnectedness, temporality and spirituality, and positiveness or expectancy. A higher score of the sum or the 3 sub scales indicates a higher hope level with scores ranging from 12 to 48.
Cancer-related Fatigue Scale (CFS) | Baseline and up to 12 weeks (post-intervention)
  An instrument consisting of 15 items that assess physical, affective, and cognitive dimensions of fatigue at present moment, with Likert scales ranging from 1 to 5. the physical sub scale consists of 7 items, the affective sub scale consists of 4 items, and the cognitive sub scale consists of 3 items and the total of all 3 sub scales indicate that greater scores correspond to greater fatigue levels.
Visual Analogue Scale for Hope (VAS-H) | obtained 6 times throughout the completion of intervention (up to 12 weeks)
  VAS is a single, frequent measurement to address the current levels of hope. Its s based on a 100cm horizontal line from 1cm (hopeless) to 100cm (hopeful)
Visual Analogue Scale for Fatigue (VAS-F) | Obtained 6 times throughout the completion of intervention (up to 12 weeks)
  VAS is a single, frequent measurement to address the current levels of fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Hannibal, PhD, Study Director — Aalborg University
Locations (1):
- Aretaieion University Hospital, Athens, Attica, Greece